CLINICAL TRIAL: NCT05055700
Title: Assessing the Impact of a Mobile App on Pregnant Women's Perceptions, Knowledge, and Uptake of Prenatal Genetic Testing
Brief Title: Impact of a Mobile App on Pregnant Women's Prenatal Genetic Testing Decision-making
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Collaborators: Driscoll Children's Hospital (Other); Global Institute for Hispanic Health (Unknown)
Responsible Party: Principal Investigator, Lei-Shih Chen, Professor, Texas A&M University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 0004459
Record Dates: First submitted 2021-09-14; First posted 2021-09-24 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Pregnant Women; Mobile Applications; Genetic Testing; Prenatal Care

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): This arm will review a mobile app to learn information about prenatal genetic testing before their appointment with maternal-fetal medicine specialists.
  Interventions: Behavioral: Mobile app with prenatal genetic testing information
- Control group (No Intervention): This arm will only receive usual care - visit maternal-fetal medicine specialists.

INTERVENTIONS:
Behavioral: Mobile app with prenatal genetic testing information — In the intervention group, participants will be asked to download, register, and review a mobile app on their own mobile phones before their appointment with maternal-fetal medicine specialists. This mobile app includes prenatal genetic testing information about amniocentesis, chorionic villus sampling, nuchal translucency screening, cell-free DNA, triple/quad/penta screening, anatomy ultrasound, and carrier screening.
  Arms: Intervention group

SUMMARY:
Determine the effect of a culturally sensitive prenatal genetic testing (PGT) education intervention delivered via a mobile application on pregnant women's perceptions, knowledge, and uptake of PGT. Our working hypothesis, based on prior studies, is that pregnant women who receive a culturally sensitive intervention to enhance their knowledge and understanding of PGT will feel more confident in their decision-making regarding PGT.

ELIGIBILITY:
Inclusion Criteria -

Women who:

1. age over 18 years old;
2. are able to speak, read and, write English or Spanish;
3. are currently pregnant;
4. have a smartphone with IOS or Android;
5. are current prenatal patients in one of the prenatal clinics in the Driscoll Health System;
6. were referred to the clinic because they are at high risk of having a baby with genetic conditions (e.g., advanced maternal age, family history, history of delivering affected baby, abnormal blood or ultrasound screening results).

Exclusion Criteria -

Women who:

1. are unable to speak, read, and write English or Spanish;
2. do not own a smartphone with IOS or Android system.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Attitudes toward prenatal genetic testing | From the time of enrollment to two weeks after the participants' appointment with maternal-fetal medicine specialists.
  Measured by a 4-item scale that asks participants how they feel about prenatal genetic testing.
Knowledge about prenatal genetic testing | From the time of enrollment to two weeks after the participants' appointment with maternal-fetal medicine specialists.
  Measured by 27 knowledge questions about prenatal genetic testing options' timing, procedures, and purposes.
Decisional conflicts about prenatal genetic testing | From the time of enrollment to two weeks after the participants' appointment with maternal-fetal medicine specialists.
  Measured by the modified 5-item SURE Decisional Conflicts scale.
Uptake of prenatal genetic testing | Within one year after the intervention.
  Participants' decisions on prenatal genetic testing by reviewing participants' medical charts.

SECONDARY OUTCOMES:
Psychological symptom [Anxiety] | From the time of enrollment to two weeks after the participants' appointment with maternal-fetal medicine specialists.
  Measured by the 6-item sub-scale of Brief Symptom Inventory-18 about anxiety.
Decision Self-Efficacy about prenatal genetic testing | From the time of enrollment to two weeks after the participants' appointment with maternal-fetal medicine specialists.
  Measured by the modified 11-item Decision Self-Efficacy scale.
Preparation for Decision Making about prenatal genetic testing | From the time of enrollment to two weeks after the participants' appointment with maternal-fetal medicine specialists.
  Measured by the modified 7-item Preparation for Decision Making scale.

CONTACTS AND LOCATIONS:
Overall Officials: Lei-Shih Chen, PhD, Principal Investigator — Texas A&M University; Robin Page, Principal Investigator — Texas A&M University
Locations (1):
- Driscoll Children's hospital, Corpus Christi, Texas, United States

IPD SHARING:
Plan to Share IPD: No